CLINICAL TRIAL: NCT02680080
Title: The Effect of Pink Grapefruit Juice on the QT Interval in Healthy Volunteers and Patients With Congenital Long QT Syndrome
Brief Title: Effect of Grapefruit on QT Interval in Healthy Volunteers and Patients With Congenital Long QT Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, michal roll, Director. Research & development, Tel-Aviv Sourasky Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-15-EC-15-0728-TLV-CTIL
Record Dates: First submitted 2016-01-28; First posted 2016-02-11 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Long QT Syndrome
MeSH Terms: conditions — Long QT Syndrome | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive control group (Active Comparator): subjects will receive a single 400 mg tablet of Moxifloxacin - the most commonly used positive control in "thorough" QTc (TQT) studies. Subjects will be continuously recorded by a Holter monitor for 24 hours
  Interventions: Drug: Moxifloxacin
- Grapefruit group (Active Comparator): subjects will drink one liter of fresh pink-grapefruit juice as fast as possible. The pink-grapefruit juice will be squeezed in the morning of the experiment in the cardiology department. ECG will be performed immediately pre dose and at 1, 2, 3, 4, 6, 8, 12, 24 after fresh pink-grapefruit juice administration. In addition, subjects will be continuously recorded by a Holter monitor for 24 hours
  Interventions: Dietary Supplement: Grapefruit group

INTERVENTIONS:
Drug: Moxifloxacin — a single 400 mg tablet of Moxifloxacin
  Arms: Positive control group
Dietary Supplement: Grapefruit group — one liter of fresh pink-grapefruit juice
  Arms: Grapefruit group

SUMMARY:
The list of medications that prolong the QT interval and can provoke torsade de pointes keeps expanding. This list includes not only antiarrhythmic drugs, but also medications with no cardiac indications. All these medications prolong the QT interval because they block a specific potassium channel on the myocardial cell membrane: the channel for the rapid component of the delayed rectifier potassium current or "IKr". The risk for developing torsade de pointes for patients taking any of the medications with IKr blockade capabilities varies from >4% for antiarrhythmic drugs to <0.01% for non-cardiac medications. The risk depends on the strength of IKr blockade, but also on specific patient characteristics. The majority of patients who develop torsade de pointes from non-cardiac medications have identifiable risk factors. In this regard, patients with a congenital long QT syndrome are prone to develop torsade de pointes when treated with QT-prolonging medications. This is because, due to their genetically defective ion channels, patients with Long QT Syndrome (LQTS) have impaired ventricular repolarization and reduced "repolarization reserve." Therefore, it is common medical practice to strongly advise patients with congenital LQTS to avoid all medications that have IKr channel blocker capabilities. it was reported that some flavonoids contained in pink-grapefruit juice block the IKr channel. These investigators also reported that drinking 1 liter of pink-grapefruit juice causes QT prolongation in healthy volunteers. The magnitude of the QT prolongation provoked by grapefruit juice was small However, drugs causing minor QT prolongation in healthy volunteers may provoke major QT prolongation in rare or sick individuals who are then at risk for developing torsade de pointes. Consequently, one could argue that, until proven otherwise, pink-grapefruit should be added to the list of "drugs" that are forbidden for patients with LQTS

DETAILED DESCRIPTION:
The list of medications that prolong the QT interval and can provoke torsade de pointes keeps expanding. This list includes not only antiarrhythmic drugs, but also medications with no cardiac indications (like several antibiotics, antihistamines or antipsychotic medications). All these medications prolong the QT interval because they block a specific potassium channel on the myocardial cell membrane: the channel for the rapid component of the delayed rectifier potassium current or "IKr". The risk for developing torsade de pointes for patients taking any of the medications with IKr blockade capabilities varies from >4% for antiarrhythmic drugs to <0.01% for non-cardiac medications. The risk depends on the strength of IKr blockade, but also on specific patient characteristics. In fact, the majority of patients who develop torsade de pointes from non-cardiac medications have identifiable risk factors. In this regard, patients with a congenital long QT syndrome (LQTS) are prone to develop torsade de pointes when treated with QT-prolonging medications. This is because, due to their genetically defective ion channels, patients with LQTS have impaired ventricular repolarization and reduced "repolarization reserve." Therefore, it is common medical practice to strongly advise patients with congenital LQTS to avoid all medications that have IKr channel blocker capabilities. Zitron et al reported that some flavonoids contained in pink-grapefruit juice block the IKr channel. These investigators also reported that drinking 1 liter of pink-grapefruit juice causes QT prolongation in healthy volunteers. The magnitude of the QT prolongation provoked by grapefruit juice was small (12.5 ± 4.2 msec). However, drugs causing minor QT prolongation in healthy volunteers may provoke major QT prolongation in rare or sick individuals who are then at risk for developing torsade de pointes. Consequently, one could argue that, until proven otherwise, pink-grapefruit should be added to the list of "drugs" that are forbidden for patients with LQTS.

This is a single center, open-label, randomized, crossover study. Subjects will be admitted to the cardiology department on the day before the first dose and will remain there until study completion. After performing a baseline electrocardiogram and baseline blood tests (Complete Blood Count, chemistry - up to 10 ml of blood) subjects will be continuously recorded by a Holter monitor for 24 hours (baseline Holter). On the next day subjects will be randomly divided into two experimental therapies (one after the other in a random order to the same group of patients

ELIGIBILITY:
Inclusion Criteria:

Inclusions Criteria - healthy volunteers

1. Healthy volunteers between 18 and <65 years of age.
2. Subjects within BMI 18.0-29.0 calculated as Weight (Kg)/Height (m)2.
3. No known history of significant neurological (including history of seizures or EEG abnormalities), renal, cardiovascular (including known structural cardiac abnormalities or hypertension), respiratory (asthma), endocrinological, gastrointestinal, hepatic or hematopoietic disease, neoplasm, psychological (marked anxiety, tension or agitation) or any other clinically significant medical disorder, which in the investigator's judgment contraindicate administration of the study medications.
4. No significant abnormalities in screening physical examination
5. No known allergy to Fluoroquinolone (Moxifloxacin)
6. Subjects must provide written informed consent to participate in the study
7. No significant abnormalities in the electrocardiogram prior to the first dosing day.

Inclusions Criteria - LQTS patients:

1. LQTS patients between 18 and <65 years of age.
2. Subjects within BMI 18.0-29.0 calculated as Weight (Kg)/Height (m)2.
3. No known history of significant neurological (including history of seizures or EEG abnormalities), renal, cardiovascular (including known structural cardiac abnormalities or hypertension), respiratory (asthma), endocrinological, gastrointestinal, hepatic or hematopoietic disease, neoplasm, psychological (marked anxiety, tension or agitation) or any other clinically significant medical disorder, which in the investigator's judgment contraindicate administration of the study medications.
4. No significant abnormalities in screening physical examination.
5. Subjects must provide written informed consent to participate in the study.

Exclusion Criteria:

Exclusions Criteria - healthy volunteers:

1. Subjects with any clinically significant abnormality upon physical examination or in the clinical laboratory test values (CBC, electrolytes, renal function and liver enzymes).
2. Subjects with a history of clinically defined GERD, peptic ulcer or any gastrointestinal surgery other than appendectomy or herniotomy, or with any gastrointestinal disorder likely to influence drug absorption, or with any history of severe gastrointestinal narrowing, or frequent nausea or emesis, regardless of etiology.
3. Subjects with significant allergic response to other drugs or history of food allergies deemed clinically significant or exclusionary for the study.
4. Previous episode of syncope or seizures.
5. Supine heart rate < 45 beats per minute after 5 minutes rest.
6. QTc prolongation (defined as QTc >450 msec for healthy volunteers) in the electrocardiogram on screening examination.
7. Significant abnormalities in the electrocardiogram prior to the first dosing day. Patients with sinus arrhythmia will be excluded.
8. Subjects with an inability to communicate well with the investigators and staff (i.e., language problem, poor mental development or impaired cerebral function).
9. Subjects with any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by the Principal Investigator.
10. Subjects who are non-cooperative or unwilling to sign consent form.

Exclusions Criteria - LQTS patients:

1. Subjects with any clinically significant abnormality upon physical examination or in the clinical laboratory test values (CBC, electrolytes, renal function and liver enzymes).
2. Subjects with a history of clinically defined GERD, peptic ulcer or any gastrointestinal surgery other than appendectomy or herniotomy, or with any gastrointestinal disorder likely to influence drug absorption, or with any history of severe gastrointestinal narrowing, or frequent nausea or emesis, regardless of etiology.
3. Subjects with significant allergic response to other drugs or history of food allergies deemed clinically significant or exclusionary for the study.
4. Previous episode of syncope or seizures.
5. Supine heart rate < 45 beats per minute after 5 minutes rest.
6. QTc prolongation (defined as QTc >500 msec for LQTS patients) in the electrocardiogram on screening examination.
7. Subjects with an inability to communicate well with the investigators and staff (i.e., language problem, poor mental development or impaired cerebral function).
8. Subjects with any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by the Principal Investigator.
9. Subjects who are non-cooperative or unwilling to sign consent form.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
QT measurements | up to 24 hours
  ECG will be performed after fresh pink-grapefruit juice administration. In addition, subjects will be continuously recorded by a Holter monitor for 24 hours QT interval, RR and QTc will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Chorin, MD, Principal Investigator — Tel Aviv MC
Locations (1):
- Sourasky medical center (Ichilov), Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chorin E, Hochstadt A, Granot Y, Khoury S, Schwartz AL, Margolis G, Barashi R, Viskin D, Ghantous E, Schnapper M, Mekori T, Fourey D, Guevara-Valdivia ME, Marquez MF, Zeltzer D, Rosso R, Viskin S. Grapefruit juice prolongs the QT interval of healthy volunteers and patients with long QT syndrome. Heart Rhythm. 2019 Aug;16(8):1141-1148. doi: 10.1016/j.hrthm.2019.04.039. Epub 2019 May 8. PMID 31075442